CLINICAL TRIAL: NCT05023109
Title: A Study to Evaluate GP Chemotherapy in Combination With Tislelizumab and Ociperlimab as First-line Treatment in Participants With Unresectable Advanced Biliary Tract Carcinoma (BTC)
Brief Title: GP Chemotherapy in Combination With Anti-PD-1 and Anti-TIGIT in Unresectable Advanced BTC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Jining Medical University (Other); Cancer Hospital of Guangxi Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZSAB-TOP
Record Dates: First submitted 2021-08-20; First posted 2021-08-26 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Biliary Tract Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GP+PD-1+Tight (Experimental): Tislelizumab 200mg IV Q3W + Ociperlimab 900mg IV Q3W + GP (gemcitabine 1000mg/m2 + cisplatin 25mg/m2 Q3W) Gemcitabine/Cisplatin will be administered on D1/D8 in every three weeks cycle and up to 8 cycles.
  Tislelizumab and Ociperlimab will be administered on D1 in every three weeks cycle, until the disease progression, intolerable toxicity, death, withdrawal of consent.
  Interventions: Drug: GP+PD-1+Tight

INTERVENTIONS:
Drug: GP+PD-1+Tight — Drug: Tislelizumab Tislelizumab 200mg IV Q3W
  Other Name:
  BGB-A317 Anti-PD-1 therapy
  Drug: Ociperlimab Ociperlimab 900mg IV Q3W
  Other Name:
  BGB-A1217 Anti-TIGIT therapy
  Drug: GP chemotherapy gemcitabine 1000mg/m2 + cisplatin 25mg/m2 Q3W

SUMMARY:
This is an open label, multi-center, phaseⅡstudy to evaluate the efficacy and safety of GP (Gemcitabine/Cisplatin) in combination with Tislelizumab and Ociperlimab as first-line treatment in participants with unresectable advanced Biliary Tract Carcinoma (BTC).

DETAILED DESCRIPTION:
Biliary Tract Carcinoma (BTC) has an insidious onset, invasiveness, high malignancy, and no specific symptoms in the early stage, and most of them are in the middle and advanced stages at the time of diagnosis and have lost the chance of surgery. For patients with advanced BTC, systemic therapy is currently the main choice, and gemcitabine/cisplatin (GP) is currently the "gold standard" for first-line treatment of advanced BTC, but the efficacy is still unsatisfactory, and more and more clinical practice has found that GP-based combination therapy may have better efficacy.

Previous studies have shown that chemotherapy can improve the immunotherapy microenvironment and may have a synergistic anti-tumor effect in combination with immunotherapy. This study is to explore the efficacy and safety of GP in combination with anti-PD1 antibody (Tislelizumab) and anti-TIGIT antibody (Ociperlimab) as first-line treatment in participants with unresectable advanced BTC.

ELIGIBILITY:
Inclusion Criteria:

* • Subjects with a histopathological or cytologically diagnosis of BTC

  * The participants must be required to sign an informed consent
  * At least one measurable lesion (RECIST 1.1)
  * No previous systematic treatment for BTC
  * Child-Pugh Score, Class A
  * ECOG performance status 0 or 1
  * Adequate organ function
  * Life expectancy of at least 3 months

Exclusion Criteria:

* • Diagnosis of mixed ampullary, hepatocellular, and cholangiocarcinoma

  * Known history of a serious allergy to any monoclonal antibody
  * Known central nervous system metastases and/or leptomeningeal disease prior to treatment
  * Portal hypertension with esophageal or gastric varices within 6 months prior to initiation of treatment
  * Any bleeding or thrombotic disorder within 6 months prior to initiation of treatment
  * Any active malignancy prior to the start of treatment
  * Active or history of autoimmune disease
  * Other acute or chronic conditions, psychiatric disorders, or laboratory abnormalities that may increase the risk of study participation
  * Pregnant or lactating women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-01-18 (Actual); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 24 months
  ORR is defined as the proportion of subjects with complete response (CR) or partial response (PR) to study drugs

SECONDARY OUTCOMES:
Disease control rate (DCR) | 24 months
  DCR is defined as the proportion of subjects with CR or PR or SD to study drugs
Duration of response (DoR) | 24 months
  DoR is defined as the time interval from first meeting response criteria (CR or PR) to confirmed progressive disease (PD) or death, whichever occurs first.
Progression-free survival (PFS) | 24 months
  PFS is defined as the time from the date of treatment to the first documented disease progression or death due to any cause, whichever occurs first.
6-months/12-months PFS rate | 6 months/12 months
  6-months/12-months PFS rate is defined as the proportion of patients alive and free of disease progression at 6 months/12 months.
Overall Survival (OS） | 24 months
  OS is defined as the time from the treatment until death due to any cause.
6-months/12-months OS rate | 6 months/12 months
  OS rate is defined as the proportion of patients who have not experienced death from any cause at 6 months/12 months.
Adverse Events (AEs) | 24 months
  The grade of AEs and the number of patients with AEs are assessed based on CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Jia Fan, Principal Investigator — Shanghai Zhongshan Hospital
Locations (1):
- Zhongshan hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No